CLINICAL TRIAL: NCT06156930
Title: Erciyes University Faculty of Health Sciences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ayser DÖNER, Research assistant (Principal Investigator), TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Erciyes University Health
Record Dates: First submitted 2023-11-16; First posted 2023-12-05 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Restless leg syndrome; Aromatherapy massage; Sleep quality; Lavender oil
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: three-armed
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group Lavander (Experimental): The group will receive aromatherapy massage with a 5% mixture prepared with sesame oil and lavender oil for 10 minutes on both lower leg areas, three times a week for four weeks.
  Interventions: Other: Intervention group lavender oil
- Placebo group sesame (Placebo Comparator): The group will receive a massage with sesame oil on both lower leg areas for 10 minutes on each leg, three times a week for four weeks.
  Interventions: Other: Placebo group sesame oil
- Control group (No Intervention): Group of individuals receiving HD treatment who do not receive any treatment other than standard treatment

INTERVENTIONS:
Other: Intervention group lavender oil — The group will receive aromatherapy massage with a 5% mixture prepared with sesame oil and lavender oil for 10 minutes on both lower leg areas, three times a week for four weeks.
  Other Names: Lavender oil aromatherapy massage
  Arms: Intervention group Lavander
Other: Placebo group sesame oil — The group will receive a massage with sesame oil on both lower leg areas for 10 minutes on each leg, three times a week for four weeks.
  Other Names: Sesame oil massage
  Arms: Placebo group sesame

SUMMARY:
Sleep disorders are important to place among the symptoms frequently seen in hemodialysis patients. Among sleep disorders, restless legs syndrome is the most common. Restless legs syndrome, seen in patients receiving hemodialysis treatment, causes excessive daytime sleepiness and negatively affects the sleep quality of individuals.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years or older,
* Not pregnant and not planning a pregnancy,
* Having been diagnosed with restless leg syndrome according to the restless leg syndrome diagnostic scale and by a physician,
* Having at least mild restless leg syndrome according to the restless leg syndrome severity rating scale,
* Scoring 11 or above on the Epworth sleepiness scale,
* PSQI score an average of 5 and above,
* Receiving hemodialysis treatment in hemodialysis units for at least 3 months and 3 sessions per week,
* Continuing dialysis treatment in the same institution,
* Able to walk independently,
* No changes in the treatment program before the massage and throughout the research process,
* Not having any allergies to the oils to be used,
* Individuals who can understand and communicate with Turkish will be included in the research

Exclusion Criteria:

* Those who are sensitive and/or have any allergies to the lavender oil to be used,
* Those who have lower leg problems that would prevent them from applying massage to the lower leg area,
* Have a history of mental or physical disability, including peripheral neuropathy, vascular problems in the legs,
* Epilepsy, Alzheimer's, Parkinson's, Multiple Sclerosis, etc. Those with a diagnosed neurological disease such as
* Pre-implemented,
* Those with respiratory system disorders,
* Patients who used other complementary and integrative therapies methods during the study period will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
RLS Severity Rating Scale | Change compared to the initial score 1 month after aromatherapy massage application
  The RLS Severity Rating Scale was developed in 2003. The scale was applied in the selection of patients and in the weekly evaluation of RLS severity. The scale comprised ten questions; each question was scored between 0 and 4. Questions 1, 2, 4, 6, 7, and 8 were related to RLS symptoms, questions 5, 9, and 10 were related to the effect of the disease on the mental state and daily social activities of patients with RLS, and question 3 was about the diagnostic criteria of RLS. The overall score indicated the RLS severity. A minimum score of 0 and a maximum score of 40 could be obtained. A score between 1 and 10 corresponded to "mild," 11-20 "moderate," 21-30 "severe," and 31-40 "very severe" RLS.
Epworth Sleepiness Scale | Change compared to the initial score 1 month after aromatherapy massage application
  Daytime sleepiness is determined with the scale developed in 1991. The scale consists of 8 questions in total and a high score from the scale indicates an increased level of daytime sleepiness. With this four-point Likert type scale, each question is rated between 0-3. In the evaluation of the scale; 0-5 points: normal, 6-10 points: normal but increased daytime sleepiness, 11-12 points: increased moderate daytime sleepiness, 13-15 points: increased moderate daytime sleepiness, 16-24 points: increased severe daytime sleepiness It is considered as sleepiness. The minimum score is 0, the maximum score is 24, and a total score of 11 or above indicates excessive daytime sleepiness of individuals.

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | Change compared to the initial score 1 month after aromatherapy massage application
  PSQI is a reliable and valid index that measures sleep quality. The total score in the PSQI, which consists of 24 items and is divided into 7 sections (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorder, use of sleeping pills and daytime dysfunction), varies between 0-21, and the PSQI total score is 5 and below. A score above 5 indicates that the sleep quality is 'good', and a score above 5 indicates that the sleep quality is 'bad'.

CONTACTS AND LOCATIONS:
Overall Officials: AYSER DÖNER, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans.

REFERENCES:
- [Background] Doner A, Tasci S. Effect of massage therapy with lavender oil on severity of restless legs syndrome and quality of life in hemodialysis patients. J Nurs Scholarsh. 2022 May;54(3):304-314. doi: 10.1111/jnu.12738. Epub 2021 Nov 14. PMID 34779137
- [Background] Ghasemi M, Rejeh N, Bahrami T, Heravi-Karimooi M, Tadrisi SD, Vaismoradi M. Aromatherapy Massage vs. Foot Reflexology on the Severity of Restless Legs Syndrome in Female Patients Undergoing Hemodialysis. Geriatrics (Basel). 2021 Oct 11;6(4):99. doi: 10.3390/geriatrics6040099. PMID 34698176
- [Background] Hashemi SH, Hajbagheri A, Aghajani M. The Effect of Massage With Lavender Oil on Restless Leg Syndrome in Hemodialysis Patients: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Dec;4(4):e29617. doi: 10.17795/nmsjournal29617. Epub 2015 Dec 1. PMID 26835466
- [Background] Malekshahi, F., Aryamanesh, F., Fallahi, S. 2018.
- [Background] Mirbagher Ajorpaz N, Rahemi Z, Aghajani M, Hashemi SH. Effects of glycerin oil and lavender oil massages on hemodialysis patients' restless legs syndrome. J Bodyw Mov Ther. 2020 Jan;24(1):88-92. doi: 10.1016/j.jbmt.2019.06.012. Epub 2019 Jun 29. PMID 31987569
- [Background] Mohammadpourhodki R, Sadeghnezhad H, Ebrahimi H, Basirinezhad MH, Maleki M, Bossola M. The Effect of Aromatherapy Massage With Lavender and Citrus Aurantium Essential Oil on Quality of Life of Patients on Chronic Hemodialysis: A Parallel Randomized Clinical Trial Study. J Pain Symptom Manage. 2021 Mar;61(3):456-463.e1. doi: 10.1016/j.jpainsymman.2020.08.032. Epub 2020 Sep 1. PMID 32889038
- [Background] Muz G, Tasci S. Effect of aromatherapy via inhalation on the sleep quality and fatigue level in people undergoing hemodialysis. Appl Nurs Res. 2017 Oct;37:28-35. doi: 10.1016/j.apnr.2017.07.004. Epub 2017 Aug 1. PMID 28985917
- [Background] Nasiri M, Abbasi M, Khosroabadi ZY, Saghafi H, Hamzeei F, Amiri MH, Yusefi H. Short-term effects of massage with olive oil on the severity of uremic restless legs syndrome: A double-blind placebo-controlled trial. Complement Ther Med. 2019 Jun;44:261-268. doi: 10.1016/j.ctim.2019.05.009. Epub 2019 May 8. PMID 31126564
- [Background] Oshvandi K, Mirzajani Letomi F, Soltanian AR, Shamsizadeh M. The effects of foot massage on hemodialysis patients' sleep quality and restless leg syndrome: a comparison of lavender and sweet orange essential oil topical application. J Complement Integr Med. 2021 Apr 12;18(4):843-850. doi: 10.1515/jcim-2020-0121. PMID 33838094
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Allen RP, Picchietti D, Hening WA, Trenkwalder C, Walters AS, Montplaisi J; Restless Legs Syndrome Diagnosis and Epidemiology workshop at the National Institutes of Health; International Restless Legs Syndrome Study Group. Restless legs syndrome: diagnostic criteria, special considerations, and epidemiology. A report from the restless legs syndrome diagnosis and epidemiology workshop at the National Institutes of Health. Sleep Med. 2003 Mar;4(2):101-19. doi: 10.1016/s1389-9457(03)00010-8. PMID 14592341
- [Background] Allen RP, Picchietti DL, Garcia-Borreguero D, Ondo WG, Walters AS, Winkelman JW, Zucconi M, Ferri R, Trenkwalder C, Lee HB; International Restless Legs Syndrome Study Group. Restless legs syndrome/Willis-Ekbom disease diagnostic criteria: updated International Restless Legs Syndrome Study Group (IRLSSG) consensus criteria--history, rationale, description, and significance. Sleep Med. 2014 Aug;15(8):860-73. doi: 10.1016/j.sleep.2014.03.025. Epub 2014 May 17. PMID 25023924
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Hening WA, Allen RP. Restless legs syndrome (RLS): the continuing development of diagnostic standards and severity measures. Sleep Med. 2003 Mar;4(2):95-7. doi: 10.1016/s1389-9457(03)00009-1. No abstract available. PMID 14592339
- [Background] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342